CLINICAL TRIAL: NCT01943981
Title: Exercise Performance in Patients With Atrial Fibrillation: Usefulness of Cardiopulmonary Exercise Test
Brief Title: Exercise Performance in Patients With Atrial Fibrillation
Acronym: AF-CPX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Mi-Jeong Kim, Assistant professor, Incheon St.Mary's Hospital
Other Study IDs: OC13OISI0099
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optimal/inappropriate exercise response

SUMMARY:
Heart failure and stroke are the two major complication of atrial fibrillation. Current treatment for atrial fibrillation is so focused to stroke prevention, but the risk assessment for heart failure is less highlighted. The most of patients with atrial fibrillation have cardiac functional limitation of variable degree. We hypothesize that the exercise test would reveal the subclinical cardiac dysfunction, and might be helpful to classify the patients with atrial fibrillation according to their exercise capacity real cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Nonvalvular chronic atrial fibrillation
* Left ventricular ejection fraction >40%

Exclusion Criteria:

* Acute decompensated heart failure within 30 days
* unstable hemodynamic status
* Significant coronary artery disease
* Any condition interfering sufficient exercise
* Valvular stenosis or regurgitation of moderate or severe degree
* Obstructive or restrictive lung disease of moderate or severe degree
* Active malignancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and preserved left ventricular systolic function
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Exercise response patterns of heart rate and oxygen uptake | At baseline

SECONDARY OUTCOMES:
Composite cardiovascular events (all death, admission of heart failure, stroke/thromboembolism) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St.Mary's Hospital, Incheon, South Korea